CLINICAL TRIAL: NCT05249322
Title: FollowMuco : Study of Satisfaction of Patients and Care Providers for an Alternate Follow-up With In-hospital Consults and Tele-consult for Patients With Cystic Fibrosis
Brief Title: Study of Satisfaction of Patients and Care Providers for an Alternate Follow-up With In-hospital Consults and Tele-consult for Patients With Cystic Fibrosis
Acronym: FollowMuco
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL21_1354; 2022-A00134-39 (Other: ID-RCB)
Record Dates: First submitted 2022-01-27; First posted 2022-02-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cystic Fibrosis
Keywords: tele-medicine; cystic fibrosis; alternate follow-up
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Follow-up alternating between face-to-face consultation and teleconsultation every three months (Experimental): Patients of this arm will be followed alternating between face-to-face consultation and teleconsultation respecting the recommended frequency (every three months) during 12 months (M+3:teleconsultation - M+6:in-hospital consultation - M+9:teleconsultation - M+12 : in-hospital consultation)
  Interventions: Other: Follow-up alternating between face-to-face consultation and teleconsultation every three months.

INTERVENTIONS:
Other: Follow-up alternating between face-to-face consultation and teleconsultation every three months. — The intervention will be an alternate follow-up every three months with:
  * A tele-consult: with paramedical consult (with assistance for home-spirometry) and medical consult for about 1h30 in total, make with a HCL platform for telemedicine.
  * An usual in-hospital consult of about 1h30 with paramedical and medical consult.

SUMMARY:
The pandemic forced us to develop home follow-up for patients with chronical diseases . In the same time, the new era of treatment for cystic fibrosis considerably improves the health of patients with this pathology.

This study aims to assess the satisfaction of patients and care providers for an alternated follow-up between tele-consults and in-hospital consults during one year for patients with cystic fibrosis treated by Kaftrio® since at least one year and stable.

ELIGIBILITY:
Inclusion Criteria:

* patients with cystic fibrosis
* Patients treated with Kaftrio® since one year
* autonomous patients
* patients without cognitive disorders
* Patients voluntary for this follow up
* patients with two tele-communication tools
* patients with FEV1>50%
* patients with less of 2 antibiotics cure per year

Exclusion Criteria:

* all transplanted patients
* Pregnant patients
* Particular follow up needed in-hospital consult
* Persons deprived of their liberty by a judicial or administrative decision
* Persons subject to psychiatric care
* Persons admitted to a health or social establishment for purposes other than research
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patients and care providers satisfaction after one year of alternated follow-up (hospital Consults and Tele-consult) | Measured at inclusion and after one year of follow up.
  Satisfaction of patients and care providers for the follow-up by the Client-Satisfaction-Questionnaire (CSQ-8 for patients and CSQ-3 for care-provider). For the CSQ-8 the minimum value is 8 and the maximum value is 32. There is three levels: Low satisfaction (8-20), medium satisfaction (21-26) and high satisfaction (27-32) .

SECONDARY OUTCOMES:
Patients and care providers satisfaction for tele consultation | Measured after tele-consult (at 6 month M+6 and at 12 month M+12)
  Satisfaction of patients and care providers for tele-consults by telemedicine satisfaction Questionnaire (TSQ).
  The TSQ is a 14-item questionnaire in its final version, the questionnaire items are scored on a five-point scale, from 1 being strongly disagree to 5 being strongly agree.. The internal consistency of the TSQ was 0.93, which is considered acceptable and indicates strong correlations between the items that make up the scale. Predictive validity supported the conclusion that the TSQ measured patient satisfaction with telemedicine (Pearson's correlation coefficient (r=0.45, P<0.05).
Comparison between FEV1 measured at the department's respiratory functional exploration center and FEV1 measured with the Spirobank ® during the same in-hospital visit. | At inclusion, 6month and 12 month
  Comparison between FEV1 measured at the department's respiratory functional exploration center and FEV1 measured with the Spirobank ® during the same in-hospital visit in order to check that the difference between the two values does not exceed the margin of error of 5%.
effect on Patients and care providers quality of life | Measured at inclusion and after one year
  Quality of life of patients by Cystic fibrosis questionnaire revised(CFQ-R). The CFQ-R is a validated patient-reported outcome measuring health-related quality of life for children and adults with CF. The CFQ-R contains both general and CF-specific scales. The CFQ-R was administered at Days 0, 14, 28, and 42. The endpoint was change in respiratory symptoms (e.g., coughing, congestion, wheezing) from Day 0 (baseline), assessed with the CFQ-R RSS (score range: 0-100; higher scores indicating fewer symptoms, higher health-related quality of life, or better functioning). Baseline CFQ-R RSS and age group (<18 vs. >=18 years) were included as covariates in the analysis.
effect on Patients FEV1 (Forced expiratory volume) | Measured at inclusion and after one year
  FEV1 measured in start and at the end of the study
effect on Patients antibiotic cure number | Measured at inclusion and after one year
  Antibiotic cure during one year before start and after one year of the study
effect on patient's weight | Measured at inclusion and after one year
  Weight measured in start and at the end of the study
Effect on Patients call and mail to CF center | Measured at inclusion and after one year
  Number of calls and mails to CF center during one year before start and after one year of the study

CONTACTS AND LOCATIONS:
Overall Officials: Thomas VIDAL, Principal Investigator — adult cystic fibrosis centre Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France